CLINICAL TRIAL: NCT04294979
Title: Study on the Interaction Between Immune, Autonomic and Central Nervous Systems as a Target of Exercise Therapy in Multiple Sclerosis
Brief Title: Exercise Therapy in Multiple Sclerosis
Acronym: RehaMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Neuromed IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 19/13
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; exercise; Multiple sclerosis; Physical therapy
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Rehabilitation (Experimental): Conventional Physical Therapy
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The rehabilitation program will consist of both passive and active therapeutic exercises specifically aimed at restoring or maintaining muscular flexibility, range of motion, balance, coordination of movements, postural passages and transfers, and ambulation. . Furthermore, advanced robotic therapy such as Lokomat® exoskeleton (Hocoma AG, Volketswil, Switzerland), Biodex® Stability System (BSS, Biodex, Inc, Shirley, NY), G-EO System™ (Reha Technology AG, Olten, Svizzera) and Indego® Therapy (Parker USA), will be used to personalize rehabilitation treatment.
  Other Names: Exercise

SUMMARY:
Exercise or active rehabilitation is a non-pharmacological approach increasingly used for people with Multiple Sclerosis (MS), in support of disease-modifying therapies (DMTs), with the aim of improving the quality of life and engagement in daily activities. Exercise improves several disease outcomes, like cardiovascular and neuromuscular functions and walking abilities. However, its disease modifying potential is poorly explored. Exercise might target two relevant disease hallmarks that are interconnected, such as the dysregulated immune system and the inflammatory synaptopathy. Exercise might act through the activation of the autonomic part of the vagus nerve, which is an important modulator of both the innate and adaptive immune system, through the so-called cholinergic anti-inflammatory pathway-CAP.

This study aims to address the effect of exercise in reducing peripheral inflammation that drives the synaptic pathology and neurodegeneration occurring in the brain of MS patients. Patients will undergo a therapeutic exercise program, consisting of 3 hours of treatment per day, 6 days/week for a total of 6 weeks. The treatment will include both passive and active therapeutic exercises targeted to restore or preserve muscular flexibility, motor coordination and ambulatory function. The day of recruitment (time 0) patients will undergo neurological and mood examination and blood withdrawal to analyze peripheral markers of immune function. Moreover, transcranial magnetic stimulation (TMS) will be used to measure synaptic transmission, while the heart rate variability (HRV) test will be performed to explore vagal function. The effect of exercise will be evaluated at the end of rehabilitation (after 6 weeks-time 1), on the above parameters. A follow up will be included (time 2, 8 weeks after the end of the treatment) to address long-term effects on neurologic and mood measurements as well as peripheral marker levels.

DETAILED DESCRIPTION:
Clinical manifestations of Multiple Sclerosis (MS) indicate the involvement of motor, sensory, visual systems, cognition and emotion, as well as peripheral autonomic system (PAS). Disease modifying therapies (DMTs) are immunomodulatory drugs designed to dampen the immune reaction occurring in MS. Indeed, MS pathogenesis is supposed to rely on the break of immunological tolerance against myelin epitopes, which trigger an inflammatory cascade that leads to chronic inflammation, axonal loss and neurodegeneration. T cell population in MS presents several metabolic dysfunctions, such as glycolysis alterations that can be attenuated by DMTs. Studies of synaptic transmission conducted on both MS patients, via transcranial magnetic stimulation (TMS), and EAE mice, via electrophysiological recordings of single neurons, showed an early synaptopathy characterized by an impairment of glutamatergic and GABAergic transmissions. Such synaptopathy is independent of demyelination and caused by inflammation. Importantly, TMS cortical excitability measures positively correlate with disability in MS patients. Moreover, chimeric experiments obtained incubating MS T cells and murine brain slices, clearly indicate that T cells drive synaptic damage during MS, suggesting that interfering with T cell-neuron crosstalk could be a possible therapeutic target.

Due to the complexity and the heterogeneity of the disease course and the clinical symptoms, the search for the appropriate personalized treatment and the disease management remains a challenging issue. It is increasingly recognized that a multi-disciplinary approach in MS treatment, including non-pharmacological interventions is required to treat MS. Active-rehabilitation or exercise has been proven effective in the improvement of cardiovascular functions, aerobic capacity, muscular strength and ambulatory performance, while some data indicate that other outcomes, like balance and depression can be positively influenced by exercise. Symptoms of sympathovagal imbalance, like altered heart rate variability (HRV), previously shown to depend on inflammatory bulk in MS, may be positively modulated by exercise, which is known to regulate both the peripheral nervous system and the immune system. However, the mechanisms involved in exercise-beneficial effects as well as the impact of exercise on MS pathophysiological hallmarks, especially those regarding the immune-synaptic axis, are still poorly elucidated.

This longitudinal, interventional, non-pharmacological study is designed to enrol 44 MS patients and 30 healthy controls matched by gender and age to the MS group. The MS patient group will undergo a conventional 6-week rehabilitation program. Physical therapy will be performed for 6 days/week for 6 weeks and will consist of 3 hours of treatment per day. The rehabilitation program will be planned by a physician specialized in physical and rehabilitation medicine and will consist of both passive and active therapeutic exercises specifically aimed at restoring or maintaining muscular flexibility, range of motion, balance, coordination of movements, postural passages and transfers, and ambulation. According to the patient's disability status, different therapeutic exercises will be performed by qualified physiotherapists. Intensity of exercise will be tailored to the level of patient's disability. Furthermore, advanced robotic therapy such as Lokomat® exoskeleton (Hocoma AG, Volketswil, Switzerland), Biodex® Stability System (BSS, Biodex, Inc, Shirley, NY), G-EO System™ (Reha Technology AG, Olten, Svizzera) and Indego® Therapy (Parker USA), will be used to standardize rehabilitation treatment and obtain more objective indices of motor function and will be applied according to clinical indications. Three time-points (t) of evaluations are included in the study: t0 (before starting the rehabilitation period), t1 (soon after rehabilitation) and t2 (follow-up, after 8 weeks by the end of rehabilitation). Therapeutic efficacy will be evaluated at the end of the exercise program (t1) by repeating evaluations performed at t0, which include neurological and psychological assessments, together with measures of brain synaptic activity and vagal function and immune function. At t2, analysis will be limited to neurological and psychological assessments and immune function. Thus, blood samples will be collected at t0, t1 and t2 to study changes in immune function that might correlate with clinical parameters described as primary and secondary outcomes at the different time-points.

Statistical analysis will be performed by IBM SPSS Statistics 15.0. Data will be tested for normality distribution through the Kolmogorov-Smirnov test. Differences between pre- and post-values will be analyzed using parametric Student's t-test for matched pairs, or if necessary, nonparametric Wilcoxon signed-rank test for matched pairs. Changes in categorical variables will be assessed by McNemar test. Correlation analysis will be performed by calculating Pearson or Spearman coefficients as appropriate. Changes in categorical variables will be evaluated by the test McNemar. Data will be presented as the mean (standard deviation, sd) or median (25th- 75th percentile). The significance level is established at p<0.05.

Sample size calculation was performed according to the following criteria. Assuming that in MS patients the cytokine values in particular the TNF level after exercise therapy decrease in a manner similar to that showed in the study by Hedegaard et al (2008). Based on these results, calculating an average difference between pre and post exercise values of TNF equal to 1365.1 pg / ml (sd = 2570), d = 0.53, in order to appreciate a moderate effect with a statistical capacity of 95% and assuming a two-tailed a = 0.05 and applying a Wilcoxon rank test for paired values, the investigators estimate a total number of patients equal to 40. Analysis was performed with the G * POWER v3.1.9.2 program. Considering possible drop-outs, the investigators estimate to increase the number of patients recruited by one percentage equal to 10%, meaning 4 subjects. Moreover, using Power Analysis d=0.61, it has been calculated that the number of healthy volunteer subjects needed to be recruited for the study of the immunophenotype and secretoma will be 30 subjects per experimental group, in order to be able to refuse the null hypothesis that the two groups are equal with a test power of 95% and appreciate a difference of 1600.9 pg / ml between the means of the experimental groups (healthy control vs MS) (standard deviation equal to 2599), d = 0.61. The probability of Type I error associated with this test for this hypothesis is 5%.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent to the study;
* Diagnosis of MS definite according to 2010 revised McDonald's criteria (Polman et al., 2011);
* Age range 18-65 (included);
* EDSS range between 4,5 and 6,5 (included);
* Ability to participate to the study protocol.

Exclusion Criteria:

* Inability to provide written informed consent to the study;
* Altered blood count;
* Female with a positive pregnancy test at baseline or having active pregnancy plans in the following months after the beginning of the protocol;
* Contraindications to gadolinium (MRI);
* Contraindications to TMS;
* Patients with comorbidities for a neurological disease other than MS, included other neurodegenerative chronic diseases or chronic infections (i.e tuberculosis, infectious hepatitis, HIV/AIDS);
* Unstable medical condition or infections;
* Use of medications with increased risk of seizures (i.e. Fampridine, 4- Aminopyridine);
* Concomitant use of drugs that may alter synaptic transmission and plasticity (cannabinoids, L-dopa, antiepileptics, nicotine, baclofen, SSRI, botulinum toxin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in clinical disability (EDSS) | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Clinical severity will be measured by the expanded disability status scale (EDSS): this scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Changes in clinical disability: Multiple Sclerosis Functional Composite (MSFC) | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  The Multiple Sclerosis Functional Composite (MSFC) is a three-part composite clinical measure that includes three variables: Timed 25-Foot walk; 9-Hole Peg Test; and Paced Auditory Serial Addition Test (PASAT-3"). The results from each of these three tests are transformed into Z-scores and averaged to generate a composite score for each patient at each time point. There are 3 components: 1. the average scores from the four trials on the 9-HPT; 2. the average scores of two 25-Foot Timed Walk trials; 3. the number correct from the PASAT-3. The scores for these three dimensions are combined to create a single score that can be used to detect variations over time, by creating Z-scores for each component. MSFC Score = {Zarm, average + Zleg, average + Zcognitive} / 3.0 (Where Zxxx =Z-score). Increased scores represent deterioration in the 9-HPT and the 25-Foot Timed Walk, whereas decreased scores represent deterioration in the PASAT-3.
Changes in visual disability | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  The visual acuity test (VA) will be performed using Snellen scales and low-contrast letter acuity (LCLA).

SECONDARY OUTCOMES:
Changes in Mood-depressive trait | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Depression level will be assessed by the Beck Depression Inventory-Second Edition (BDI-II) (Watson et al, 2014), a self-administered questionnaire of 21 items.
Changes in Mood-anxiety trait | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  The level of anxiety will be assessed by State-Trait Anxiety Inventory (STAI) form Y (STAI-Y), a 40-item self-administered questionnaire measuring anxiety as a state (situational anxiety) or trait (long-standing propensity to anxious mood).
Neurophysiological assessment | Changes from baseline (time 0, t0) to the end of the 6-week exercise protocol (time 1, t1)
  Cortical excitability will be measured with TMS using Magstim stimulators (Magstim Company, UK) to an eight-shaped coil placed tangentially on the scalp to elicit motor evoked potentials (MEP) in the first dorsal interosseous muscle of the dominant hand. The motor thresholds will be calculated at rest (RMT) as the lowest stimulus intensity capable of evoking a MEP of about 50 uV in five out of ten stimuli, and during a slight voluntary contraction of the target muscle as the minimum intensity capable of evoking MEP> 100 uV in five out of ten stimuli. To test the interhemispheric inhibition (IHI) a double pulse TMS paradigm will be applied. Long term potentiation (LTP) will be evaluated using the intermittent theta-burst stimulation protocol (iTBS). iTBS consists of a three pulses train delivered at the frequency of 50 Hz and repeated every 200 ms for a total of 600 stimuli, with an intensity equal to 80% of the AMT at the M1 of the dominant hemisphere.
Changes in autonomic function | Changes from baseline (time 0, t0) to the end of the 6-week exercise protocol (time 1, t1)
  Heart rate variability (HRV) will be measured through standard procedures. The analysis of ECG (ET Medical Devices SpA) will be performed in the frequency domain using dedicated software (Light-SNV software). The periods heart rate (HR) lasting 5 minutes will be chosen from the last 6 minutes of supine rest lasting 30 minutes. The spectral power analysis will consider an ad component high frequency (HF) (0.16-0.4 Hz), which mainly reflects vagal activity, and a low component frequency (LF) (0.04-0.15 Hz), which mainly reflects sympathetic activity. The will be considered spectral components in normalized units (LFnu, HFnu). The LF / HF ratio will be used as an index of sympathetic-vagal balance.
Changes in T cell function | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Immediately after collection in Vacutainer tubes containing anticoagulant, peripheral blood samples, will be processed for isolation of T lymphocytes by centrifugation according to standardized techniques, and frozen at -80 in the shortest possible time. T cells isolated will be analyzed at flow cytometer to analyze the phenotype and cell subpopulations, after staining for surface antigens (CD3, CD4, CD8, CD25, CD28, CD45RA, CD69, CD71, CCR7) and intracellular labelling for specific cytokines (IFN-g, TNFa, IL-2, IL-17, IL-4). A portion of these cells will be cultured to evaluate their secretome (cytokines) via ELISA / Luminex assay and cellular metabolism via SeaHorse assay. Data will be expressed as picograms per milliliter (pg/ml) (ELISA/Lumiex assay) and extracellular acidification rate-ECAR- in mpH/min (Seahorse assay).
Electrophysiological evaluation | Changes from baseline (time 0, t0), to the end of the 6-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  T lymphocytes will be used for performing chimeric experiments based on T cell incubation with murine corticostriatal and hippocampal slices to measure glutamatergic transmission and LTP, respectively, using techniques of single neuron electrophysiology on murine brain slices.

CONTACTS AND LOCATIONS:
Overall Officials: Antonietta Gentile, phD, Principal Investigator — IRCCS San Raffele Pisana
Locations (1):
- IRCCS San Raffele Pisana, Roma, RM, Italy

REFERENCES:
- [Background] Mandolesi G, Gentile A, Musella A, Fresegna D, De Vito F, Bullitta S, Sepman H, Marfia GA, Centonze D. Synaptopathy connects inflammation and neurodegeneration in multiple sclerosis. Nat Rev Neurol. 2015 Dec;11(12):711-24. doi: 10.1038/nrneurol.2015.222. Epub 2015 Nov 20. PMID 26585978
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890
- [Background] Charron S, McKay KA, Tremlett H. Physical activity and disability outcomes in multiple sclerosis: A systematic review (2011-2016). Mult Scler Relat Disord. 2018 Feb;20:169-177. doi: 10.1016/j.msard.2018.01.021. Epub 2018 Feb 2. PMID 29414293
- [Background] Gentile A, De Vito F, Fresegna D, Rizzo FR, Bullitta S, Guadalupi L, Vanni V, Buttari F, Stampanoni Bassi M, Leuti A, Chiurchiu V, Marfia GA, Mandolesi G, Centonze D, Musella A. Peripheral T cells from multiple sclerosis patients trigger synaptotoxic alterations in central neurons. Neuropathol Appl Neurobiol. 2020 Feb;46(2):160-170. doi: 10.1111/nan.12569. Epub 2019 Jun 17. PMID 31125471
- [Background] Carbone F, De Rosa V, Carrieri PB, Montella S, Bruzzese D, Porcellini A, Procaccini C, La Cava A, Matarese G. Regulatory T cell proliferative potential is impaired in human autoimmune disease. Nat Med. 2014 Jan;20(1):69-74. doi: 10.1038/nm.3411. Epub 2013 Dec 8. PMID 24317118
- [Background] Feys P, Giovannoni G, Dijsselbloem N, Centonze D, Eelen P, Lykke Andersen S. The importance of a multi-disciplinary perspective and patient activation programmes in MS management. Mult Scler. 2016 Aug;22(2 Suppl):34-46. doi: 10.1177/1352458516650741. PMID 27465614
- [Background] Hedegaard CJ, Krakauer M, Bendtzen K, Sorensen PS, Sellebjerg F, Nielsen CH. The effect of beta-interferon therapy on myelin basic protein-elicited CD4+ T cell proliferation and cytokine production in multiple sclerosis. Clin Immunol. 2008 Oct;129(1):80-9. doi: 10.1016/j.clim.2008.06.007. Epub 2008 Jul 23. PMID 18653385
- [Background] Lanzillo R, Carbone F, Quarantelli M, Bruzzese D, Carotenuto A, De Rosa V, Colamatteo A, Micillo T, De Luca Picione C, Sacca F, De Rosa A, Moccia M, Brescia Morra V, Matarese G. Immunometabolic profiling of patients with multiple sclerosis identifies new biomarkers to predict disease activity during treatment with interferon beta-1a. Clin Immunol. 2017 Oct;183:249-253. doi: 10.1016/j.clim.2017.08.011. Epub 2017 Aug 18. PMID 28823971
- [Background] La Rocca C, Carbone F, De Rosa V, Colamatteo A, Galgani M, Perna F, Lanzillo R, Brescia Morra V, Orefice G, Cerillo I, Florio C, Maniscalco GT, Salvetti M, Centonze D, Uccelli A, Longobardi S, Visconti A, Matarese G. Immunometabolic profiling of T cells from patients with relapsing-remitting multiple sclerosis reveals an impairment in glycolysis and mitochondrial respiration. Metabolism. 2017 Dec;77:39-46. doi: 10.1016/j.metabol.2017.08.011. Epub 2017 Sep 8. PMID 29132538
- [Background] Pavlov VA, Tracey KJ. Neural regulation of immunity: molecular mechanisms and clinical translation. Nat Neurosci. 2017 Feb;20(2):156-166. doi: 10.1038/nn.4477. Epub 2017 Jan 16. PMID 28092663
- [Background] Studer V, Rocchi C, Motta C, Lauretti B, Perugini J, Brambilla L, Pareja-Gutierrez L, Camera G, Barbieri FR, Marfia GA, Centonze D, Rossi S. Heart rate variability is differentially altered in multiple sclerosis: implications for acute, worsening and progressive disability. Mult Scler J Exp Transl Clin. 2017 Apr 5;3(2):2055217317701317. doi: 10.1177/2055217317701317. eCollection 2017 Apr-Jun. PMID 28607756
- [Background] Mori F, Kusayanagi H, Monteleone F, Moscatelli A, Nicoletti CG, Bernardi G, Centonze D. Short interval intracortical facilitation correlates with the degree of disability in multiple sclerosis. Brain Stimul. 2013 Jan;6(1):67-71. doi: 10.1016/j.brs.2012.02.001. Epub 2012 Feb 24. PMID 22425067
- [Background] Mori F, Kusayanagi H, Nicoletti CG, Weiss S, Marciani MG, Centonze D. Cortical plasticity predicts recovery from relapse in multiple sclerosis. Mult Scler. 2014 Apr;20(4):451-7. doi: 10.1177/1352458513512541. Epub 2013 Nov 21. PMID 24263385
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Background] Sternberg Z. Promoting sympathovagal balance in multiple sclerosis; pharmacological, non-pharmacological, and surgical strategies. Autoimmun Rev. 2016 Feb;15(2):113-23. doi: 10.1016/j.autrev.2015.04.012. Epub 2015 May 3. PMID 25945428
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Centonze D, Muzio L, Rossi S, Cavasinni F, De Chiara V, Bergami A, Musella A, D'Amelio M, Cavallucci V, Martorana A, Bergamaschi A, Cencioni MT, Diamantini A, Butti E, Comi G, Bernardi G, Cecconi F, Battistini L, Furlan R, Martino G. Inflammation triggers synaptic alteration and degeneration in experimental autoimmune encephalomyelitis. J Neurosci. 2009 Mar 18;29(11):3442-52. doi: 10.1523/JNEUROSCI.5804-08.2009. PMID 19295150
- [Background] Gentile A, Musella A, De Vito F, Rizzo FR, Fresegna D, Bullitta S, Vanni V, Guadalupi L, Stampanoni Bassi M, Buttari F, Centonze D, Mandolesi G. Immunomodulatory Effects of Exercise in Experimental Multiple Sclerosis. Front Immunol. 2019 Sep 13;10:2197. doi: 10.3389/fimmu.2019.02197. eCollection 2019. PMID 31572399
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Schulz KH, Gold SM, Witte J, Bartsch K, Lang UE, Hellweg R, Reer R, Braumann KM, Heesen C. Impact of aerobic training on immune-endocrine parameters, neurotrophic factors, quality of life and coordinative function in multiple sclerosis. J Neurol Sci. 2004 Oct 15;225(1-2):11-8. doi: 10.1016/j.jns.2004.06.009. PMID 15465080